CLINICAL TRIAL: NCT00936286
Title: The Impact of Respiratory Muscle Training on the Therapy of Obstructive Sleep Apnea Syndrome (OSAS) Patients
Brief Title: Respiratory Muscle Training in Obstructive Sleep Apnea Syndrome (OSAS) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Idiag AG (Industry)
Responsible Party: Prof. Dr. med. Winfried J. Randerath, Wissenschaftliches Institut Bethanien e.V.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WI_SpiroTiger_87/2008
Record Dates: First submitted 2009-07-07; First posted 2009-07-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Obstructive Sleep Apnea Syndrome; Respiratory Muscle Training; Normocapnic Hyperpnea; SpiroTiger; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Respiratory Muscle Training (Experimental)
  Interventions: Device: SpiroTiger

INTERVENTIONS:
Device: SpiroTiger — Respiratory muscle training with SpiroTiger device, 1 week training initiation and 4 weeks training period with 5 training days per week, training duration 30 min each. Respiratory bag volume set at 50% VC, respiratory frequency starting from 50% MVV. Weekly control trainings.
  Other Names: SpiroTiger Medical

SUMMARY:
The purpose of this study is to determine whether respiratory muscle training by means of normocapnic hyperpnea leads to clinical and polysomnographical improvements in patients with mild to intermediate sleep apnea syndrome.

DETAILED DESCRIPTION:
The obstructive sleep apnea syndrome (OSAS) is of great significance for affected individuals as well as for public health service. Patients suffer from reduced quality of life and show an increased accident risk in road traffic and on the job. Furthermore, OSAS represents an independent risk factor for cardiovascular diseases, in particular arterial hypertension.

In sleep apnea patients, the relatively early stimulation of the upper respiratory tract muscles compared to the thoracic respiratory muscles is abrogated in many cases. Alternatively, nerve damage with impaired sensory function in the pharynx area and impaired motor function of the upper air tract musculature, in particular the musculus genioglossus can be observed. The disturbed sensory function impairs the reflex activation of the genioglossus. Moreover, the pattern of neurogenic muscle damage with a loss of the pattern of different types of fibers changed to the point of adjoining atrophic and hypertrophic sections and a more monotonous appearance of fiber types could be detected. During waking hours the activity of the musculus genioglossus is enhanced compared with control persons, which is interpreted as a compensatory mechanism. During sleep time, however, this compensation seems to disappear.

In several studies either direct or indirect stimulation of the musculus genioglossus and its supplying nerves were deployed. Yet, the results were inconsistent. The direct muscle stimulation using intramuscular electrodes, although efficient, was no longer pursued due to technical reasons. Although the results of an external stimulation showed improvements regarding apneas and snoring, the findings were usually weakly pronounced. In a study ascertaining muscle training with transcutaneous electrical stimulation a significant improvement regarding snoring was achieved when compared to placebo. In general, no influence on sleep apnea syndrome could be accomplished, although there were individual cases showing a clinically relevant amelioration.

A preceding study compared habitual snorers with control persons. It was shown that respiratory muscle training by means of normocapnic hyperpnea was accompanied by enlargement of the musculus genioglossus and reduced snoring. Moreover, an increased physical performance was observed.

Thus, the question arises if training of the respiratory musculature by means of normocapnic hyperpnea leads to clinical and polysomnographical improvements in patients with mild to intermediate sleep apnea syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Mild to intermediate sleep apnea syndrome with AHI of 10 - 30/h and clinical symptoms
* Refusal of a primary nCPAP therapy
* Epworth Sleepiness Scale (ESS) score ≥ 9
* Signed informed consent form

Exclusion Criteria:

* Therapy with pharmaceuticals which can influence the musculature
* Psychiatric disease which negatively influences compliance
* Acute and chronic diseases of the lung and/or the respiratory passages
* BMI ≥ 35 kg/m²

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index, Snoring | 5 weeks

SECONDARY OUTCOMES:
Polysomnography (PSG) with sleep stages, total arousal count and respiratory arousal count | 5 weeks
Clinical symptoms according to self-assessment questionnaire (Epworth Sleepiness Scale) | 5 weeks
Lung function test parameters (VC, FEV1, MVV, etc.) | 5 weeks
Nocturnal partial pressure of oxygen and/or carbon dioxide in the blood (during PSG) | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Winfried J. Randerath, Prof. Dr., Study Chair — Wissenschaftliches Institut Bethanien e.V
Locations (1):
- Wissenschaftliches Institut Bethanien e.V., Solingen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Herkenrath SD, Treml M, Priegnitz C, Galetke W, Randerath WJ. Effects of respiratory muscle training (RMT) in patients with mild to moderate obstructive sleep apnea (OSA). Sleep Breath. 2018 May;22(2):323-328. doi: 10.1007/s11325-017-1582-6. Epub 2017 Oct 28. PMID 29080065